CLINICAL TRIAL: NCT01724476
Title: A Placebo-Controlled Trial of Folate With B12 in Patients With Schizophrenia With Residual Symptoms in Ethiopia
Brief Title: A Trial of Folate With B12 in Patients With Schizophrenia With Residual Symptoms in Ethiopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Addis Ababa University (Other); Amanuel Mental Hospital, Addis Ababa, Ethiopia (Unknown)
Responsible Party: Principal Investigator, Gregory Fricchione, Director, Chester M. Pierce, MD Division of Global Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011P002667; 2011D003142 (Other: InfoEd proposal number)
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folate with B12 (Active Comparator): Subjects randomized to the folate with B12 group will take 1 capsule of 400mcg per day of folate with B12.
  Interventions: Drug: folate with B12
- placebo (Placebo Comparator): Subjects randomized to the placebo group will take 1 capsule of placebo per day.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: folate with B12
  Arms: folate with B12
Drug: placebo
  Arms: placebo

SUMMARY:
The investigators propose to conduct a randomized Sequential Parallel Design for Double-Blind Phase fixed dose, 4-month trial of folate plus B12 as add-on therapy in 200 Ethiopian subjects with schizophrenia with stable residual positive or negative symptoms.

DETAILED DESCRIPTION:
This is a 16-week, randomized, double-blind, placebo-controlled study of Folate 2mg plus B12 400mcg, as an adjunctive therapy in approximately 240 consecutive outpatients with schizophrenia from Amanuel Hospital, which is based at Addis Ababa, Ethiopia will be enrolled and screened for eligibility. The goal is to randomize and complete 200 subjects from the 240 enrolled. A Sequential Parallel Design for Double-Blind Phase will be utilized. During the first phase of double-blind adjunctive treatment, eligible patients (n=200) are randomized to adjunctive treatment with either folate and vitamin B12 (n=60) or placebo (n=150), with a 2:3:3 ratio for random assignment to the treatment sequences drug/drug (DD; n=70), placebo/placebo (PP; n=70), and placebo/drug (PD; n=75), while all continue to receive their antipsychotic agent for the entire duration of the study. Assuming a 10% drop-out rate during the first phase, 126 patients on placebo will complete the first 56-day phase, and 54 patients on folate and vitamin B12 will complete the first 56-day phase.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, any subtype
2. Male or female
3. Age 18-65 years
4. Treated with an antipsychotic for at least 6 months at a stable dose for at least 6 weeks
5. PANSS total score of at least 60, with at least a 3 (moderate) on one negative symptom item or on one positive symptom item.
6. No acute medical problems; any chronic medical condition (e.g. hypertension) consistently treated and stable during the 1 month prior to participation

Exclusion Criteria:

1. Unable to provide informed consent
2. Serum B12 concentration less than 300mcg/L; Complete Blood Count (CBC) results consistent with megaloblastic anemia
3. Serum creatinine concentration greater than 1.4
4. Current use of folate or B12 supplementation
5. Current use of any of the following medications: phenobarbital, phenytoin, carbamazepine, valproic acid, fosphenytoin, primidone or pyrimethamine; antimalarial drugs
6. Alcohol or other substance abuse within 3 months (nicotine allowed)
7. Subjects with a history of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders (e.g. unstable angina, decompensated congestive heart failure, Central Nervous System (CNS) infection or history of HIV seropositivity), which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study. Active medical conditions that are minor or well controlled are not exclusionary if they do not affect risk to the patient or the study results. For example, the following are not exclusionary: a) stable and well- controlled hypertension; b) asthma (no serious attacks in the past year)
8. Unstable psychiatric illness
9. Seizure disorder
10. Pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of schizophrenia as measured by the change from baseline in Positive and Negative Syndrome Scale (PANSS) total score | Baseline to Week 16
  Examine the efficacy of a four-month trial of folate supplementation with B12 for potentially reducing symptoms of schizophrenia as measured by the change from baseline in Positive and Negative Syndrome Scale (PANSS) total score

SECONDARY OUTCOMES:
Change in psychotic symptoms as measured by the PANSS psychosis subscale score | Baseline to Week 16
  Examine the efficacy of folate supplementation with B12 for psychotic symptoms as measured by the PANSS psychosis subscale score
Change in negative symptoms as measured by the Scale for Assessment of Negative Symptoms (SANS) | Baseline to Week 16
  Examine the efficacy of folate supplementation with B12 for negative symptoms as measured by the modified Scale for Assessment of Negative Symptoms (SANS) total score

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Fricchione, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Amanuel Mental Hospital, Addis Ababa, Ethiopia